CLINICAL TRIAL: NCT01562704
Title: Visualisation of the Central Analgesic Effect of Paracetamol in Functional MRI
Acronym: IRMf
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Dr. Gisèle PICKERING (MCU, PH) (Unknown); Dr. Betty JEAN (PH) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0110
Record Dates: First submitted 2012-01-27; First posted 2012-03-26 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Pain
Keywords: mechanism of action of paracetamol in the brain structures
MeSH Terms: conditions — Pain | interventions — Acetaminophen; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- paracetamol (Experimental)
  Interventions: Drug: Paracetamol (drug)
- placebo (Placebo Comparator)

INTERVENTIONS:
Drug: Paracetamol (drug) — The objective of this study is to evaluate the mechanism of action of paracetamol (versus placebo) in the brain with new assessment tools (functional MRI and test inducing pain by thermal stimulation
  Arms: paracetamol

SUMMARY:
Paracetamol is one of the most widely used analgesic in the world, indicated for the symptomatic treatment of fever and pain. The objective of this study is to evaluate the mechanism of action of paracetamol (versus placebo) in the brain with new assessment tools (functional MRI and test inducing pain by thermal stimulation.

DETAILED DESCRIPTION:
Visit 1 / Visit 2 Inclusion of the subject, Clinical examination Trainings tests

Study period 1 Clinical examination Measurement of the basal pain thresholds Administration of product (T0) T0+100min : Thermal stimulation according to the established paradigm and fMRI data acquisition T0+180min : Thermal stimulation according to the established paradigm and fMRI data acquisition

Study period 2: same of period 1.

ELIGIBILITY:
Inclusion Criteria:

* - Healthy volunteers
* Aged at last 18 years and over 60 years
* Male
* Non-smoking subject
* Fasting coffe, tea, coca-cola or other stimulant products since the last evening
* Subject free of any treatment within 7 days prior to inclusion including no use of analgesics or anti-inflammatory treatments

Exclusion Criteria:

* Contraindications to the administration of paracetamol
* Contraindications to the completion of MRI
* Medical history and/or surgical judged by the investigator as being incompatible with the test
* Progressive disease at the inclusion

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Difference between the matrice plans obtained in both treatments (paracetamol or placebo) and 100 min after administration of paracetamol or placebo in brain structures | 100 min after administration of paracetamol or placebo

SECONDARY OUTCOMES:
Difference between the matrice plans obtained in both treatments (paracetamol or placebo) and 180 min after administration of paracetamol or placebo in brain structures | 180 min after administration of paracetamol or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Pickering G, Kastler A, Macian N, Pereira B, Valabregue R, Lehericy S, Boyer L, Dubray C, Jean B. The brain signature of paracetamol in healthy volunteers: a double-blind randomized trial. Drug Des Devel Ther. 2015 Jul 23;9:3853-62. doi: 10.2147/DDDT.S81004. eCollection 2015. PMID 26229445